CLINICAL TRIAL: NCT03120026
Title: A Whey Protein-based Nutritional Supplement Enriched in Vitamin D, Leucine and Calcium for Sarcopenia in Older Adults Undergoing Physical Rehabilitation the IRIS (Improving Rehabilitation In Sarcopenia) Study: a Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: Improving Rehabilitation In Sarcopenia (IRIS)
Acronym: IRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Principal Investigator, Mariangela Rondanelli, Principal Investigator, Azienda di Servizi alla Persona di Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20170011726
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Product (Experimental): Two servings (40 grams each) of powder (Fortifit; Nutricia) which has to be dissolved in 125 ml of water. Per serving, 20 g whey protein, 3 g total leucine, 9 g carbohydrates, 3 g fat, 800 IU vitamin D, and a mixture of vitamins, minerals, and fibers.
  Interventions: Dietary Supplement: Experimental product
- Isocaloric Placebo (Placebo Comparator): Two servings (40 grams each) of an isocaloric (maltodextrins) powder which has to be dissolved in 125 ml of water.
  Interventions: Dietary Supplement: Isocaloric placebo

INTERVENTIONS:
Dietary Supplement: Experimental product — Two servings (40 grams each) of powder (Fortifit; Nutricia) which has to be dissolved in 125 ml of water. Per serving, 20 g whey protein, 3 g total leucine, 9 g carbohydrates, 3 g fat, 800 IU vitamin D, and a mixture of vitamins, minerals, and fibers.
  Arms: Experimental Product
Dietary Supplement: Isocaloric placebo — Two servings (40 grams each) of an isocaloric (maltodextrins) powder which has to be dissolved in 125 ml of water.
  Arms: Isocaloric Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled supplementation trial tested the hypothesis that nutritional supplementation with muscle-target nutritional supplementation concurrent with regular, controlled physical activity would increase the efficacy of physical rehabilitation in old adults suffering from sarcopenia

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled supplementation trial tested the hypothesis that nutritional supplementation with whey protein, essential amino acids - mainly leucine - vitamin D and calcium concurrent with regular, controlled physical activity would increase the efficacy of physical rehabilitation in old adults suffering from sarcopenia

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* admission for physical rehabilitation
* sarcopenia, measured with bioelectrical impedance assessment (BIA) + handgrip strength and gait speed
* Mini Mental State Examination ≥18
* Informed consent

Exclusion Criteria:

* Any malignant disease during the last five years
* Known kidney failure (previous glomerular filtration rate <30 ml/min);
* Known liver failure (Child B or C)
* Psychiatric disease
* Endocrine disorders associated with disorders of calcium metabolism (excluding osteoporosis)
* Indications related to the study product:

More than 10 µg (400 IU) of daily Vitamin D intake from medical sources More than 500 mg of daily calcium intake from medical sources. Adherence to a high energy or high protein diet up or use of protein containing or amino acid containing nutritional supplements up to three months before starting the study.

* Known allergy to milk, milk products or other components of the proposed interventions
* Indication to or ongoing artificial nutrition support
* Inclusion in other nutrition intervention trials
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* Refusal

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Gait speed | 8 weeks
  Change in gait speed (4-meter walking test)/month

SECONDARY OUTCOMES:
Physical performance - Tinetti | 8 weeks
  Change in Tinetti scale
Physical performance - Timed Up and Go test | 8 weeks
  Change in timed up and go test
Physical performance - chair-stand | 8 weeks
  chair-stand test
Functional status - Barthel | 8 weeks
  Change in Barthel index score
Functional status - ADL | 8 weeks
  Change in activities of daily living (ADL) score
Functional status - handgrip strength | 8 weeks
  Change in handgrip strength
Body weight | 8 weeks
  Change in body weight
Muscle mass | 8 weeks
  Change in appendicular muscle mass
Cognitive function - trail making test | 8 weeks
  Change in trail making test
Cognitive function - Mini Mental State Examination | 8 weeks
  Change in Mini Mental State Examination
Quality of life | 8 weeks
  Change in 12-item Short-Form Health Survey score (physical/mental components)
Costs | 8 weeks
  Difference in costs of care (using lenght of stay and duration of rehabilitation as surrogate measures)
Adverse events | 8 weeks
  Difference in rate of adverse events related to gastrointestinal intolerance

OTHER OUTCOMES:
Intensity of care | 8 weeks
  Reduction in the level of intensity of care on a ordinal scale
Type of discharge | 8 weeks
  Proportion of patients discharged at home

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Rondanelli, MD, PhD, Study Director — Azienda di Servizi alla Persona di Pavia
Locations (2):
- Italy (2):
  - Geriatric physical medicine and rehabilitation division at the Istituto Santa Margherita - Azienda di Servizi alla Persona di Pavia, Pavia
  - Geriatric physical medicine and rehabilitation division at the Istituto Santa Margherita, Azienda di Servizi alla Persona di Pavia, Pavia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rondanelli M, Cereda E, Klersy C, Faliva MA, Peroni G, Nichetti M, Gasparri C, Iannello G, Spadaccini D, Infantino V, Caccialanza R, Perna S. Improving rehabilitation in sarcopenia: a randomized-controlled trial utilizing a muscle-targeted food for special medical purposes. J Cachexia Sarcopenia Muscle. 2020 Dec;11(6):1535-1547. doi: 10.1002/jcsm.12532. Epub 2020 Sep 22. PMID 32961041